CLINICAL TRIAL: NCT03660202
Title: A Prospective Multicenter Single-arm Clinical Trial Assessing the Safety and Effectiveness of Firesorb Sirolimus Target Eluting Bioresorbable Vascular Scaffold for the Treatment of Coronary Artery Disease: FUTURE III
Brief Title: Trial for MicroPort's Firesorb BVS: FUTURE-III
Acronym: FUTURE-III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUTURE-III
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease
Keywords: Bioresorbable Vascular Scaffold
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single Arm Safety and Effectiveness Confirmatory Study of Firesorb BVS
  Interventions: Device: Firesorb

INTERVENTIONS:
Device: Firesorb — Implantation of Sirolimus Target Eluting Bioresorbable Vascular Scaffold （Firesorb）

SUMMARY:
The FUTURE-III study is a confirmative clinical trial for Sirolimus Target Eluting Bioresorbable Vascular Scaffold (Firesorb) after the feasibility and safety of the device has been preliminary confirmed in a small-scale First-in-Man clinical trial.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single-arm trial in patients with coronary artery disease caused by up to two de novo native coronary artery lesions in separate epicardial vessels. The goal is to evaluate the safety and effectiveness of Firesorb to support the approval of the Chinese Food and Drug Administration (CFDA) for this product.All subjects will undergo clinical follow-up at 1-month, 6-month, 1-year, 2-year, 3-year, 4-year and 5-year post-index procedure. A total of 1200 subjects will be recruited, including 96 with long lesion (the scaffold to be used with a length of 33mm or 38mm) and 215 in the experimantal group of FUTURE-II clinical trial.

ELIGIBILITY:
General Inclusion Criteria:

1. 18-75 years of age, males or non-pregnant females;
2. With silent ischemia evidence, patients with stable or unstable angina, or in patients with old myocardial infarction;
3. Patients with indications for coronary artery bypass graft surgery; To understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

Angiographic Inclusion Criteria:

1. General Specification Subgroup:

   1. One or two de novo target lesions:

   If two target lesions are present, they must be present in different epicardial vessels and both must satisfy the angiographic eligibility criteria.

   Note: The definition of epicardial vessels means the LAD, LCX and RCA and their branches. Thus, the patient must not have lesions requiring treatment in e.g. both the LAD and a diagonal branch.

   b. Target lesion(s) must be located in a native coronary artery with a visually estimated stenosis ≥ 70% or ≥ 50% and < 100% with clinical evidence of myocardial ischemia, a thrombolysis in myocardial infarction (TIMI) flow of ≥1. Target lesion vessel length ≤25mm by visual estimation, target vessel diameter 2.5mm-4.0mm.

   c. Each target lesion may be covered with one stent.
2. Long Lesion Subgroup:

   1. One de novo target lesion.
   2. Target lesion(s) must be located in a native coronary artery with a visually estimated stenosis ≥ 70% or ≥ 50% and < 100% with clinical evidence of myocardial ischemia, a thrombolysis in myocardial infarction (TIMI) flow of ≥1. Target lesion vessel length ≤34mm by visual estimation, target vessel diameter 3.0mm-4.0mm.
   3. Each target lesion may be covered with one stent.

General Exclusion Criteria:

1. Within 1 week of any acute myocardial infarction or myocardial enzymes did not return to normal;
2. Implantation of stent in target vessel within 1 year;
3. Patients with planned intervention again within six months;
4. Severe congestive heart failure (NYHA III and above) ,or left ventricular ejection fraction <40% (ultrasound or left ventricular angiography);
5. Preoperative renal function serum creatinine >2.0mg/DL; receiving hemodialysis;
6. Bleeding, active gastrointestinal ulcers, brain hemorrhage or subarachnoid hemorrhage and half year history of ischemic stroke, antiplatelet agents and would not allow an anticoagulant therapy contraindications patients undergoing antithrombotic therapy;
7. Aspirin, clopidogrel, heparin, contrast agent, poly lactic acid polymer and rapamycin allergies;
8. The patient's life expectancy is less than 12 months;
9. Top participated in other drug or medical device and does not meet the primary study endpoint in clinical trials time frame;
10. Researchers determine patient compliance is poor, unable to complete the study in accordance with the requirements;
11. Heart transplantation patients;
12. The unstable arrhythmia, such as high risk ventricular extrasystole and ventricular tachycardia;
13. Cancer need chemotherapy;
14. Immunosuppression and autoimmune diseases, planned or undergoing immunosuppressive therapy;
15. Planning or being receiving long-term anticoagulant therapy, such as heparin, warfarin, etc;
16. Within six months for elective surgery requires stopping aspirin, Clopidogrel patients;
17. Blood test prompted platelet counts of less than 100x10E9/L or greater than 700x10E9/L, white blood cells than 3x10E9/L; known or suspected liver disease (such as hepatitis);
18. Peripheral vascular disease, 6F catheter is not available.

Angiographic Exclusion Criteria:

1. Left main coronary artery disease;
2. Severe triple vessel lesion and required revascularization.

The following exclusion criteria apply to the target lesion(s) or target vessel(s):

1. Aorto-ostial right coronary artery (RCA) lesion (within 3 mm of the ostium).
2. Lesion located within 3 mm of the origin of the Left Anterior Descending Artery (LAD) or left circumflex artery (LCX).
3. Lesion involving a bifurcation with a:

(1)side branch ≥ 2.5 mm in diameter, or (2)side branch with diameter stenosis ≥ 50%, or (3)side branch requiring guide wire, or (4)side branch requiring dilatation. 4. Anatomy proximal to or within the lesion that may impair delivery of Firesorb :

1. Extreme angulation (≥ 90°) proximal to or within the target lesion.
2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
3. Moderate or heavy calcification proximal to or within the target lesion. 5. Lesion or vessel involves a myocardial bridge. 6. Vessel contains thrombus as indicated in the angiographic images or by IVUS or OCT.

7. Vessel has been previously treated with a stent at any time prior to the index procedure such that the Firesorb or XIENCE would need to cross the stent to reach the target lesion.

8. Vessel has been previously treated and the target lesion is within 5 mm proximal or distal to a previously treated lesion.

9. Lesion which prevents successful balloon pre-dilatation, defined as full balloon expansion with the following outcomes:

1. Residual %DS is a maximum of < 40% (per visual estimation), ≤ 20% is strongly recommended.
2. TIMI Grade-3 flow (per visual estimation).
3. No angiographic complications (e.g. distal embolization, side branch closure).
4. No dissections National Heart Lung and Blood Institute (NHLBI) grade D-F.
5. No chest pain lasting > 5 minutes.
6. No ST depression or elevation lasting > 5 minutes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
The number and rate of Target Lesion Failure(TLF) | 1 year after index procedure
  Target Lesion Failure is defined as the composited endpoints of cardiac death,target vessel myocardial infarction and ischemia-driven target lesion revascularization.

SECONDARY OUTCOMES:
The number and rate of Acute Success-Device Success | From the start of index procedure to end of index procedure
  Successful delivery and deployment of the assigned scaffold at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold residual stenosis of less than 30% by visual.
Acute Success-Procedural Success | At time of procedure up to 7 days in hospital
  Achievement of final in-scaffold residual stenosis of less than 30% by visual estimation with successful delivery and deployment of at least one assigned scaffold at the intended target lesion and successful withdrawal of the delivery system for the target lesion without the occurrence of cardiac death, target vessel MI or repeat TLR.
Device-oriented composite endpoints (Target Lesion Failure) | 1 month,6 months,2 years,3 years,4 years and 5 years after index procedure
  Target Lesion Failure is defined as the composited endpoints of cardiac death,target vessel myocardial infarction and ischemia-driven target lesion revascularization.
Patient-oriented clinical composite endpoint (PoCE) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Patient-oriented clinical composite endpoint is defined as all cause death, all myocardial infarction, and any revascularization.
Death (Cardiac, Vascular, Non-cardiovascular) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment. Non-cardiovascular death: Any death not covered by the above definitions, such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
The number and rate of Myocardial Infarction (MI) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Attributable to target vessel (TV-MI), Not attributable to target vessel (NTV-MI)
The number and rate of Target Vessel Revascularization (TVR) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Ischemia-driven TVR (ID-TVR), Not ischemia-driven TVR (NID-TVR)
The number and rate of Target Lesion Revascularization (TLR) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Ischemia-driven TLR (ID-TLR), Not ischemia-driven TLR (NID-TLR)
The number and rate of Any Revascularization | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Ischemia-driven , Not ischemia-driven
The number and rate of Scaffold Thrombosis (per ARC definition) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Timing (acute, sub-acute, late and very late) Evidence (Definite and Probable)
  Timing (acute, sub-acute, late and very late) Evidence (Definite and Probable)
  Timing (acute, sub-acute, late and very late), Evidence (Definite and Probable)

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Wai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jiang J, Li C, Chen D, Song L, Cui Z, Li P, Gan L, Chen Y, Li H, Jia S, He S, Lu W, Gao R, Wang J; FUTURE III Investigators. Firesorb bioresorbable scaffold for de novo coronary artery disease: 1-year clinical outcomes. BMC Med. 2025 Jul 9;23(1):419. doi: 10.1186/s12916-025-04254-0. PMID 40629329